CLINICAL TRIAL: NCT03812419
Title: The Effect of Esomeprazole Versus Pantoprazole on Serum Cyclosporine Levels and Renal Function in Stable Kidney Transplant Recipients: A Randomized Clinical Trial
Brief Title: Esomeprazole or Pantoprazole in Renal Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Collaborators: Ain Shams University (Other); Nasser Institute For Research and Treatment (Other Government)
Responsible Party: Principal Investigator, Doaa Mohamed Salah ElDin Diab ELBohy, lecturer assisstant, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 7-2015/22
Record Dates: First submitted 2019-01-12; First posted 2019-01-23 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Kidney Transplant; Complications
Keywords: Allograft rejection; cyclosporine; kidney transplantation; proton pump inhibitors; gastric complications.
MeSH Terms: interventions — Esomeprazole; Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group I (Active Comparator): Esomeprazole 40 mg capsules once daily for 6 months
  Interventions: Drug: Esomeprazole 40 mg
- group II (Active Comparator): Pantoprazole 40 mg tablets once daily for 6 months
  Interventions: Drug: Pantoprazole 40mg

INTERVENTIONS:
Drug: Esomeprazole 40 mg — Esomeprazole 40 mg In addition, the immunosuppressant combination of CsA (Sandimmune; Novartis, East Hanover, NJ, USA), MMF (Cellcept; Roche, Basel, Switzerland) and the corticosteroid prednisolone (Solupred; Sanofi Aventis, Tours, France).
  Other Names: Ezogast
  Arms: group I
Drug: Pantoprazole 40mg — Pantoprazole 40 mg In addition, the immunosuppressant combination of CsA (Sandimmune; Novartis, East Hanover, NJ, USA), MMF (Cellcept; Roche, Basel, Switzerland) and the corticosteroid prednisolone (Solupred; Sanofi Aventis, Tours, France).
  Other Names: Pantoprazole
  Arms: group II

SUMMARY:
prospective, parallel, open-label clinical trial was performed on forty-seven adult renal transplant recipients receiving immunosuppressive therapy with CsA doses adjusted to attain trough concentrations of 100-150 μg/L, mycophenolate mofetil (MMF) at 750 mg q12 hr and prednisolone at 5 mg daily randomized into two groups, which received esomeprazole or pantoprazole at the same dose (40 mg once daily). To compare the influence of pantoprazole and esomeprazole on serum cyclosporine (CsA) levels in stable renal transplant recipients.Cyclosporine (C0), renal function and complete blood count were measured at baseline and for 6 months. Main outcome measures Clinical signs of rejection and renal function decline, assessed by serum creatinine elevations, caused by CsA level variations in either of the study groups.

DETAILED DESCRIPTION:
Study design and settings: This study is a prospective, single-centre, randomized, parallel, open-label 1:1 consecutive clinical trial of renal transplant recipients, with a follow-up 6 months; the study included an esomeprazole group (n = 25 at study completion) and a pantoprazole group (n = 22 at study completion). The study was conducted in the renal transplantation unit of the Nasser Institute in Cairo, Egypt.

Eighty renal transplant recipients were screened for eligibility. The sample size was determined by a power calculation using G power software version 3.0.10; the selected sample size showed an actual power of 0.95, α = 0.5 and an effect size of 0.8 for C0 levels of CsA and an actual power of 0.95, α = 0.5 and an effect size of 0.44 for serum creatinine levels.The participants were randomly assigned to one of two groups by single randomization. Each group received PPI therapy with a 40 mg/day dose of either esomeprazole (Ezogast; Copad Pharma, Cairo, Egypt) in group I (n = 25 at study completion) or pantoprazole (Pantoprazole; Pharo Pharma, Alexandria, Egypt) in group II (n = 22 at study completion).

In addition, participants continued to receive the immunosuppressant combination of CsA (Sandimmune; Novartis, East Hanover, NJ, USA), MMF (Cellcept; Roche, Basel, Switzerland) and the corticosteroid prednisolone (Solupred; Sanofi Aventis, Tours, France).

Administration: CsA was administered in two divided doses adjusted to achieve a C0 of 100-150 µg/L according to the transplantation centre protocol for maintenance blood CsA levels. The morning was dose separated from PPIs by at least 15 minutes, with MMF administered at 750 mg q12 hr and prednisolone administered at 5 mg daily. Each group received 40 mg/day PPI therapy on an empty stomach, and all medications were taken orally.

Renal function tests Included Parameter Assay Kits Serum creatinine QuantiChrom creatinine assay kit Blood urea nitrogen QuantiChrom urea assay kit Serum uric acid QuantiChrom uric acid assay kit Complete blood count measurements included Parameter Assay Kits Haemoglobin White blood cells (WBCs) UniCel DxH 800 Coulter Cellular Analysis System Platelets

Whole-blood C0 values in morning samples were determined spectrophotometrically using the CEDIA Cyclosporine PLUS Assay and the Indiko Plus Benchtop Analyzer (Thermo Fisher Scientific, Waltham, MA, USA)

ELIGIBILITY:
Inclusion Criteria:

* stable adult renal transplant recipients
* participants continued the same maintenance triple immunosuppressive therapy,
* triple immunosuppressive therapy was received for at least 3 years prior to the study
* transplanted 5 years before the start of the study

Exclusion Criteria:

* Paediatric patients
* patients > 65 years old
* multi-organ transplant recipients
* pregnant or lactating patients
* patients with malignancies,
* patients with active infection or inflammation
* pre-transplant GI tract disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2016-12-10 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Serum CsA (C0) level | up to 30 weeks from date of randomization untill date of any documented change in the serum concentration
  trough CsA serum levels in µg/L

SECONDARY OUTCOMES:
Serum creatinine | up to 30 weeks from date of randomization untill date of any documented change in the serum concentration
  serum creatinine concentration in mg/dl

OTHER OUTCOMES:
number of participants with signs of rejection | up to 30 weeks from date of randomization untill date of any documented rejectionoccurence of
  Fever , falnk pain , anuria

CONTACTS AND LOCATIONS:
Overall Officials: Doaa MS ElBohy, M.Sc, Principal Investigator — Future University in Egypt

IPD SHARING:
Plan to Share IPD: No